CLINICAL TRIAL: NCT02699086
Title: A Phase II Tolerability and Efficacy Study of PDC-1421 Treatment in Adult Patients With Attention-Deficit Hyperactivity Disorder (ADHD), Part I
Brief Title: A Study of PDC-1421 Treatment in Adult Patients With Attention-Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioLite, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Phase II BLI-1008-001
Record Dates: First submitted 2016-03-01; First posted 2016-03-04 (Estimated); Results first posted 2021-11-05 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Attention-Deficit Hyperactivity Disorder (ADHD)
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low dose + Low dose (Experimental): 1 PDC-1421 Capsule, trice daily, p.o. after meal for 28 + 28 days
  Interventions: Drug: PDC-1421 Capsule
- Low dose + High dose (Experimental): 1 PDC-1421 Capsule for 28 days + 2 PDC-1421 Capsules for 28 days, trice daily, p.o. after meals
  Interventions: Drug: PDC-1421 Capsule

INTERVENTIONS:
Drug: PDC-1421 Capsule — PDC-1421 Capsule is a botanical investigational new drug containing the extract of Radix Polygalae (Polygala tenuifolia Willd.) as active ingredient.

SUMMARY:
The primary objective of this trial was to determine the effective doses and treatment period of PDC-1421 Capsule in subjects with ADHD.

The secondary objective was to evaluate the safety of PDC-1421 Capsule in subjects receiving PDC-1421 at various dose levels.

DETAILED DESCRIPTION:
This study was a Part I of Phase II study designed to evaluate the safety and efficacy in adult patients with ADHD. The Screening phase is intended for diagnosing and assessing the patient for possible inclusion in the study and for providing an adequate washout period. The targeted population of this Part I study is six subjects who met the intent-to-treat per-protocol basis.

Part I study is an open-label study, single-center, and dose escalation evaluation in six patients.

1. Low dose: Six subjects will be initially evaluated for safety and efficacy assessments at low-dose (1 PDC-1421capsule TID) for 28 days. The subject will return for visit once a week during the treatment period.
2. Checkpoint #1: There will be an evaluation with all safety assessments data to decide whether subjects pass the checkpoint to enter high-dose treatment or continue to receive a low-dose treatment by the investigator.
3. High dose: The subjects who pass Checkpoint #1 will be initially evaluated for safety and efficacy assessments at high-dose (2 PDC-1421 capsules TID) for 28 days. Subjects will return for visit biweekly during the treatment period.
4. Checkpoint #2: There will be an evaluation with all safety assessments data to decide whether this study passes the checkpoint to enter Part II by the investigators.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years
2. Female subjects of child-bearing potential must test negative to pregnancy and use appropriate birth control method from the beginning of study to the 15 days later after ending of study
3. Subjects must be able to understand and willing to sign informed consent
4. Able to discontinue the use of any psychotropic medications for the treatment of ADHD symptoms at screening
5. Meet strict operational criteria for adult ADHD according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5)
6. A total score of 20 or higher on the 18-item total ADHD symptoms score of Conners' Adult Attention-Deficit/Hyperactivity Disorder Rating Scale-Self Report: Short Version (CAARS-S:S) at screening
7. Have a moderate or severe symptom of ADHD with score of 4 or higher in Clinical Global Impression-ADHD-Severity (CGI-ADHD-S) at screening

Exclusion Criteria:

1. Have any clinically significant concurrent medical condition (endocrine, renal, respiratory, cardiovascular, hematological, immunological, cerebrovascular, neurological, anorexia, obesity or malignancy) that has become unstable and may interfere with the interpretation of safety and efficacy evaluations
2. Have any clinically significant abnormal laboratory, vital sign, physical examination, or electrocardiogram (ECG) findings at screening that, in the opinion of the investigator, may interfere with the interpretation of safety or efficacy evaluations
3. Have known serological evidence of human immunodeficiency virus (HIV) antibody
4. Are pregnant as confirmed by a positive pregnancy test at screening
5. Have QTc values >450 msec at screening using Fridericia's QTc formula
6. Have current of bipolar and psychotic disorders
7. Have a current major depression disorder, obsessive-compulsive disorder, post-traumatic stress disorder, generalized anxiety disorder, panic disorder and eating disorder (also if treated but not currently symptomatic)
8. Have any history of a significant suicide attempt, or possess a current risk of attempting suicide, in the investigator's opinion, based on clinical interview and responses provided on the Beck Scale for Suicidal Ideation (BSS)
9. Have a history of jailing or imprisonment in the past 6 months due to worsening of symptoms of ADHD

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith R McBurnett, PhD, Study Director — University of California San Francisco, School of Medicine
Locations (1):
- UCSF Medical Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Dose + Low Dose | Low Dose + High Dose
Started | 0 | 6
Completed | 0 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT
Arm/Group | Low Dose + High Dose
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 38.0 [29 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Median (Full Range); unit: cm] | 178.80 [155.4 to 182.8]
Weight [Median (Full Range); unit: lb] | 170.0 [106.0 to 190.0]
ADHD Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The ADHD Rating Scale-IV with Adult Prompts is an 18-item scale base on the DSM-IV-TR criteria for ADHD that provides a rating of the severity of symptoms. The adult prompts serve as a guide to explore more fully the extent and severity of ADHD symptoms and create a framework to ascertain impairment. The odd-numbered 9 items assess inattentive symptoms and the even-numbered 9 items assess hyperactive-impulsive symptoms. Scoring is based on a 4-point, yielding a possible total score of 0-54. Higher values represent a worse outcome.
  units on a scale | 41.8 (6.6)
CAARS-S:S ADHD Index (T-score) [Mean (Standard Deviation); unit: T-scale] — Conners' ADHD Rating Scale-Self Report: Short Version (CAARS-S:S) consists of 26 Four subscales each composed of 5 items (A: inattention/memory problems; B: hyperactivity/restlessness; C: impulsivity/emotional lability; and D: problems with self-concept) as well as a 12-item ADHD index can be computed. The raw scores were converted into standard T-scores (HigherT-scores represent a worse outcome). A T-score is a standard score with a mean of 50 and a standard deviation of 10 in all samples and across all scales.
  T-scale | 73.5 (8.3)
CGI-severity [Mean (Standard Deviation); unit: score on a scale] — The Clinical Global Impression-Severity (CGI-S) is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients). CGI-I scores range from 1 (very much improved) through to 7 (very much worse).
  score on a scale | 5.3 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement ≥ 40% in ADHD-RS-IV From Baseline up to 8 Weeks Treatment
Description: The primary endpoint is the change of ADHD Rating Scale-IV (ADHD-RS-IV) total score from baseline up to Week 8 of treatment in ITT population.
  The ADHD-RS-IV with Adult Prompts is an 18-item scale base on the DSM-IV-TR criteria for ADHD that provides a rating of the severity of symptoms. The adult prompts serve as a guide to explore more fully the extent and severity of ADHD symptoms and create a framework to ascertain impairment. The odd-numbered 9 items assess inattentive symptoms and the even-numbered 9 items assess hyperactive-impulsive symptoms. Scoring is based on a 4-point, yielding a possible total score of 0-54. Likert-type severity scale: 0 = Never or Rarely, 1 = Sometimes, 2 = Often, 3 = Very Often. Clinicians should score the highest score that is generated for the prompts for each item. The ADHD-RS-IV was assessed from Visit 1 to Visit 8 by the investigator.
Time Frame: 8 weeks
Population: ITT population
Measure: Count of Participants; unit: Participants
Groups:
- Low Dose + High Dose (at Week 8): 1 PDC-1421 Capsule for 28 days + 2 PDC-1421 Capsules for 28 days, trice daily, p.o. after meals
  PDC-1421 Capsule: PDC-1421 Capsule is a botanical investigational new drug containing the extract of Radix Polygalae (Polygala tenuifolia Willd.) as active ingredient.
Arm/Group | Low Dose + High Dose (at Week 8)
Number analyzed (Participants) | 6
Participants | 5

2. Secondary Outcome: Change in ITT Population From Baseline up to 4 and 8 Weeks Treatment in the Conners' Adult Attention-Deficit/Hyperactivity Disorder Rating Scale-Self Report: Short Version (CAARS-S:S) 5 Subscales T-score.
Description: Conners' Adult Attention-Deficit/Hyperactivity Disorder Rating Scale-Self Report: Short Version (CAARS-S:S) consists of 26 items rated from 0=not at all, never to 3=very much, very frequently. Four subscales each composed of 5 items (A: inattention/memory problems; B: hyperactivity/restlessness; C: impulsivity/emotional lability; and D: problems with self-concept) as well as a 12-item ADHD index can be computed. The raw scores were converted into standard T-scores by the SAS program which was designed according to the Profile form of CAARS QuikScore forms. The higher T-scores represent a better or worse outcome. A T-score is a standard score with a mean of 50 and a standard deviation of 10 in all samples and across all scales.
Time Frame: 8 weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- Low Dose + High Dose (Week 0-4): 1 PDC-1421 Capsule for 28 days + 2 PDC-1421 Capsules for 28 days, trice daily, p.o. after meals
  PDC-1421 Capsule: PDC-1421 Capsule is a botanical investigational new drug containing the extract of Radix Polygalae (Polygala tenuifolia Willd.) as active ingredient.
  The score change is calculated from the score of week 4 comparing to week 0.
- Low Dose + High Dose (Week 0-8): 1 PDC-1421 Capsule for 28 days + 2 PDC-1421 Capsules for 28 days, trice daily, p.o. after meals
  PDC-1421 Capsule: PDC-1421 Capsule is a botanical investigational new drug containing the extract of Radix Polygalae (Polygala tenuifolia Willd.) as active ingredient.
  The score change is calculated from the score of week 8 comparing to week 0.
Arm/Group | Low Dose + High Dose (Week 0-4) | Low Dose + High Dose (Week 0-8)
Number analyzed (Participants) | 6 | 6
T-score
  Inattention/memory subscale | -10.0 (10.2) | -10.5 (11.0)
  Hyperactivity subscale | -6.2 (7.1) | -5.2 (5.9)
  Impulsivity subscale | -10.8 (7.1) | -15.2 (7.9)
  Self-concept subscale | -5.7 (7.0) | -4.7 (6.2)
  ADHD index subscale | -8.2 (7.4) | -10.8 (6.2)

3. Secondary Outcome: Number of Participants With a CGI Score of 2 or Lower
Description: Clinical Global Impression-Severity (CGI-S) and Clinical Global Impression-Improvement (CGI-I) score of 2 or lower.
  The CGI-S is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients). CGI-I scores range from 1 (very much improved) through to 7 (very much worse).
Time Frame: 8 weeks
Population: ITT population
Measure: Count of Participants; unit: Participants
Groups:
- Low Dose + High Dose (at Week 4); Low Dose + High Dose (at Week 8): 1 PDC-1421 Capsule for 28 days + 2 PDC-1421 Capsules for 28 days, trice daily, p.o. after meals
  PDC-1421 Capsule: PDC-1421 Capsule is a botanical investigational new drug containing the extract of Radix Polygalae (Polygala tenuifolia Willd.) as active ingredient.
Arm/Group | Low Dose + High Dose (at Week 4) | Low Dose + High Dose (at Week 8)
Number analyzed (Participants) | 6 | 6
Participants
  CGI-S | 0 | 2
  CGI-I | 1 | 6

4. Secondary Outcome: Change in ITT Population From Baseline up to 4 and 8 Weeks in the ADHD-RS-IV Inattention Subscale, Hyperactivity-impulsivity Subscale, and Total Scale Raw Score.
Description: The ADHD-RS-IV with Adult Prompts is an 18-item scale base on the DSM-IV-TR criteria for ADHD that provides a rating of the severity of symptoms. The adult prompts serve as a guide to explore more fully the extent and severity of ADHD symptoms and create a framework to ascertain impairment. The odd-numbered 9 items assess inattentive symptoms and the even-numbered 9 items assess hyperactive-impulsive symptoms. Scoring is based on a 4-point, yielding a possible summed "total score" of 0-54, "inattentive subscore" of 0-27, and "hyperactive-impulsive subscore" of 0-27. The higher values represent a worse outcome for the total score and subscore. Likert-type severity scale: 0 = Never or Rarely, 1 = Sometimes, 2 = Often, 3 = Very Often. . The ADHD-RS-IV was assessed from Visit 1 to Visit 8 by the investigator.
Time Frame: 8 Weeks
Population: ITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Dose + High Dose (Week 0-4) | Low Dose + High Dose (Week 0-8)
Number analyzed (Participants) | 6 | 6
score on a scale
  Inattention subscale | -10.5 (8.2) | -12.2 (7.9)
  Hyperactivity-impulsivity subscale | -7.2 (5.3) | -10.5 (4.1)
  Total scale | -17.7 (13.2) | -25.7 (11.0)

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | Low Dose + High Dose
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose + High Dose (N=6)
Eye pruritus (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Coating in mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Lethargy (General disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Irritable bowel syndrome (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/86/NCT02699086/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT02699086/SAP_001.pdf